CLINICAL TRIAL: NCT05240417
Title: Effectiveness of "Pontic-shield" Technique in Alveolar Ridge Preservation: A Randomized Controlled Trial
Brief Title: "Pontic-shield" Technique in Alveolar Ridge Preservation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jesús Torres García Denche, Associate professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21/028-EC_X
Record Dates: First submitted 2022-01-23; First posted 2022-02-15 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Tooth Extraction Status Nos; Bone Loss; Bone Resorption
Keywords: Tooth extraction; Alveolar ridge preservation; Partial extraction therapies; Bone resorption
MeSH Terms: conditions — Bone Diseases, Metabolic; Bone Resorption

STUDY DESIGN:
Intervention Model Description: Parallel three-arm randomized clinical study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group (Experimental): "Pontic-shield" will be performed as ridge preservation technique.
  Interventions: Procedure: "Pontic-shield" technique
- Positive control (ridge preservation) (Active Comparator): Deproteinized bovine bone and porcine collagen membrane will be placed after tooth extraction.
  Interventions: Procedure: Alveolar ridge preservation
- Negative control (fresh socket) (No Intervention): No intervention will be performed after tooth extraction. Blood clot will be maintained after extraction.

INTERVENTIONS:
Procedure: "Pontic-shield" technique — A 1mm thick fragment of the vestibular aspect of the root will remain after extraction (partial extraction)
  Other Names: Partial extraction therapy
  Arms: Study group
Procedure: Alveolar ridge preservation — Particulate deproteinized bovine bone and porcine collagen membrane will be placed after tooth extraction
  Arms: Positive control (ridge preservation)

SUMMARY:
Alveolar bone resorption after dental extraction frequently leads to situations in which long-term function and esthetic success of rehabilitations with dental implants is a challenge. "Pontic-shield" has been described as an alternative technique to maintain alveolar ridge after tooth extraction.

The aim of this study is to analyze the effectiveness of "Pontic-shield" technique in alveolar ridge preservation comparing to fresh socket and ridge preservation using deproteinized bovine bone and a porcine collagen membrane.

DETAILED DESCRIPTION:
A three-arm randomized clinical study will be conducted:

* Group 1 (study group): Ridge preservation with "Pontic-shield" technique.
* Group 2 (positive control): Ridge preservation with deproteinized bovine bone and porcine collagen membrane after tooth extraction.
* Group 3 (negative control): Tooth extraction only (fresh socket).

A cone-beam computed tomography will be performed prior to tooth extraction and 4 months postoperative. Radiographic changes between before and after intervention will be evaluated to asses the effectiveness of "Pontic-shield" technique.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 18 to 80 years old
* Patients who sign the informed consent
* Need to perform extraction from second premolar to second premolar in maxilla and mandible

Exclusion Criteria:

* Tobacco consumption (more than 10 cigarettes per day)
* Severe systemic disease ( ASA III or IV - American Society of Anaesthesiology)
* Drug use that could interfere with alveolar bone healing
* Active periodontal disease
* Acute or chronic apical pathology of the tooth

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Bone resorption | From the day of the extraction to 4 months after
  Radiographic changes between preoperative (prior to tooth extraction) and postoperative (4 months after intervention) will be analyzed.
  This variation will be assessed by measuring changes in width and height (in millimeters) of the socket by superimposition of CBCT before and after the intervention.

SECONDARY OUTCOMES:
Satisfaction assessed by visual analogue scale (VAS) | From the day of the surgical procedure to the seventh-day
  Postoperative pain with visual analogue scale (VAS) from 0 (no pain) to 10 (maximum pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Luis Miguel Sáez-Alcaide, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Background] Canullo L, Del Fabbro M, Khijmatgar S, Panda S, Ravida A, Tommasato G, Sculean A, Pesce P. Dimensional and histomorphometric evaluation of biomaterials used for alveolar ridge preservation: a systematic review and network meta-analysis. Clin Oral Investig. 2022 Jan;26(1):141-158. doi: 10.1007/s00784-021-04248-1. Epub 2021 Nov 26. PMID 34826029
- [Background] Saez-Alcaide LM, Gonzalez Fernandez-Tresguerres F, Cortes-Breton Brinkmann J, Segura-Mori L, Iglesias-Velazquez O, Perez-Gonzalez F, Lopez-Pintor RM, Torres Garcia-Denche J. Socket shield technique: A systematic review of human studies. Ann Anat. 2021 Nov;238:151779. doi: 10.1016/j.aanat.2021.151779. Epub 2021 Jun 1. PMID 34087383
- [Background] Hurzeler MB, Zuhr O, Schupbach P, Rebele SF, Emmanouilidis N, Fickl S. The socket-shield technique: a proof-of-principle report. J Clin Periodontol. 2010 Sep;37(9):855-62. doi: 10.1111/j.1600-051X.2010.01595.x. PMID 20712701
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354